CLINICAL TRIAL: NCT00777452
Title: A Prospective Quality of Life Study in Men With Clinically Localized Prostate Carcinoma Treated With Different Treatment Modalities
Brief Title: A Prospective Longitudinal Study of Health-Related Quality of Life in Men With Clinically Localized Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Choi Han Yong, Samsung Medical Center,Sungkyunkwan University School of Medicine
Other Study IDs: SMC IRB 2004-05-21; CRS104-10-4
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-10

CONDITIONS: Prostate Cancer
Keywords: quality of life; localized prostate cancer; FACT-P
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: active surveillance
- 2: radical prostatectomy
- 3: external beam radiotherapy
- 4: high intensity focused ultrasound

SUMMARY:
to prospectively assess the health-related quality of life (HRQOL) changes during the first year after different treatment modalities for localized prostate cancer.

DETAILED DESCRIPTION:
Quality of life is of great concern to patients considering treatment options for prostate cancer. Patients with clinically localized prostate cancer treated with active surveillance, radical prostatectomy, external radiotherapy and high intensity focused ultrasound were included. All men completed the questionnaires of Functional Assessment of Cancer Therapy-Prostate (FACT-P) (version 4), International Prostate Symptom Score (IPSS) and International Index of Erectile Function (IIEF) before treatment and 1, 3, 6, 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with clinically localized prostate cancer

Exclusion Criteria:

* patients with another malignancies

Ages: 43 Years to 82 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with clinically localized prostate cancer at single tertiary institution
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life changes over time | 12 months after treatment

SECONDARY OUTCOMES:
urinary symptom score and erectile function over time | 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Han Yong Choi, professor, Principal Investigator — Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Department of Urology, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Hashine K, Kusuhara Y, Miura N, Shirato A, Sumiyoshi Y, Kataoka M. A prospective longitudinal study comparing a radical retropubic prostatectomy and permanent prostate brachytherapy regarding the health-related quality of life for localized prostate cancer. Jpn J Clin Oncol. 2008 Jul;38(7):480-5. doi: 10.1093/jjco/hyn059. Epub 2008 Jul 11. PMID 18621847
- [Result] Namiki S, Satoh T, Baba S, Ishiyama H, Hayakawa K, Saito S, Arai Y. Quality of life after brachytherapy or radical prostatectomy for localized prostate cancer: a prospective longitudinal study. Urology. 2006 Dec;68(6):1230-6. doi: 10.1016/j.urology.2006.08.1093. Epub 2006 Dec 4. PMID 17141839
- [Result] Jo Y, Junichi H, Tomohiro F, Yoshinari I, Masato F. Radical prostatectomy versus high-dose rate brachytherapy for prostate cancer: effects on health-related quality of life. BJU Int. 2005 Jul;96(1):43-7. doi: 10.1111/j.1464-410X.2005.05564.x. PMID 15963118